CLINICAL TRIAL: NCT04705324
Title: Dilation and Curettage Versus Operative Hysteroscopy for Missed Abortion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Principal Investigator, Eli Sprecher, MD, Deputy Director Research & Development, Tel-Aviv Sourasky Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0087-20-TLV
Record Dates: First submitted 2021-01-10; First posted 2021-01-12 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Spontaneous Abortion; Missed Abortion; Intrauterine Adhesion; Retained Products of Conception
MeSH Terms: conditions — Abortion, Spontaneous; Abortion, Missed; Gynatresia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Operative Hysteroscopy (Experimental): Hysteroscopic separation
  Interventions: Procedure: Operative Hysteroscopy
- Dilation and Curettage (Active Comparator): Curettage separation
  Interventions: Procedure: D&C
- Feasibility and safety (Experimental): The first 15 patients recruited will not undergo randomization and will compose the preliminary safety and feasibility phase
  Interventions: Procedure: Operative Hysteroscopy - safety and feasibility

INTERVENTIONS:
Procedure: Operative Hysteroscopy — Separation of the non-viable gestational sac from the uterine wall will through operative hysteroscopy
  Arms: Operative Hysteroscopy
Procedure: D&C — Separation of the non-viable gestational sac from the uterine wall through dilation and curettage
  Arms: Dilation and Curettage
Procedure: Operative Hysteroscopy - safety and feasibility — Operative hysteroscopy - safety and feasibility phase
  Arms: Feasibility and safety

SUMMARY:
Randomizedtrial comparing success and complication rates of operative hysteroscopy versus traditional dilation and curettage (D&C) in the management of first trimester missed abortion.

DETAILED DESCRIPTION:
A randomized controlled trial (RCT) of women diagnosed with first trimester spontaneous abortion. Participants interested in operative evacuation of the uterus will be randomized to either operative hysteroscopy or dilation an curettage (D&C). Study population will include pregnant women diagnosed with first trimester spontaneous abortion of up to 13+0 weeks from last menstrual period (LMP) or up to 11+0 weeks of gestation as determined by Crown-Rump Length (CRL). Women who will electively choose to terminate their pregnancy as well as women diagnosed with threatened, incomplete or inevitable abortion will be excluded. All participants will undergo diagnostic hysteroscopy 6-8 weeks after allocated treatment in order to rule out intrauterine adhesion formation and retained product of conception. The primary outcome measure is the risk of intrauterine adhesion formation.

ELIGIBILITY:
Inclusion Criteria:

* Women diagnosed with missed abortion who choose to undergo surgical evacuation. and who are at gestational age of 5+0 weeks to 11+0 weeks from last menstrual period (LMP).

Exclusion Criteria:

* women who electively choose to terminate pregnancy
* women who took medical treatment for missed abortion prior to recruitment
* women with known uterine abnormality

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 55 (Estimated)
Dates: Start 2022-01-21 (Actual); Primary Completion 2024-01-20 (Estimated); Study Completion 2024-01-20 (Estimated)

PRIMARY OUTCOMES:
Intrauterine adhesions (IUA) | 2 months
  IUA formation will be assessed in all participants in the follow up diagnostic hysteroscopy performed 8 weeks after the primary treatment. IUA will be classified according to the American Society for Reproductive Medicine

SECONDARY OUTCOMES:
Retained product of conception (RPOC) | 2 months
  RPOC rate in repeat ultrasound scan performed 8 weeks after primary treatment

CONTACTS AND LOCATIONS:
Overall Officials: Yariv Yogev, M.D., Study Chair — Tel-Aviv Sourasky Medical Center
Locations (1):
- Lis Maternity Hospital, Tel Aviv Sourasky Medical Center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: Yes
Study protocol and statistical analysis plan
Supporting Information: Study Protocol, SAP
Time Frame: within 6 months of completion
Access Criteria: Yes

REFERENCES:
- [Background] Nybo Andersen AM, Wohlfahrt J, Christens P, Olsen J, Melbye M. Maternal age and fetal loss: population based register linkage study. BMJ. 2000 Jun 24;320(7251):1708-12. doi: 10.1136/bmj.320.7251.1708. PMID 10864550
- [Background] Wang X, Chen C, Wang L, Chen D, Guang W, French J. Conception, early pregnancy loss, and time to clinical pregnancy: a population-based prospective study. Fertil Steril. 2003 Mar;79(3):577-84. doi: 10.1016/s0015-0282(02)04694-0. PMID 12620443
- [Background] American College of Obstetricians and Gynecologists' Committee on Practice Bulletins-Gynecology. ACOG Practice Bulletin No. 200: Early Pregnancy Loss. Obstet Gynecol. 2018 Nov;132(5):e197-e207. doi: 10.1097/AOG.0000000000002899. PMID 30157093
- [Background] Zhang J, Gilles JM, Barnhart K, Creinin MD, Westhoff C, Frederick MM; National Institute of Child Health Human Development (NICHD) Management of Early Pregnancy Failure Trial. A comparison of medical management with misoprostol and surgical management for early pregnancy failure. N Engl J Med. 2005 Aug 25;353(8):761-9. doi: 10.1056/NEJMoa044064. PMID 16120856
- [Background] Hooker AB, Lemmers M, Thurkow AL, Heymans MW, Opmeer BC, Brolmann HA, Mol BW, Huirne JA. Systematic review and meta-analysis of intrauterine adhesions after miscarriage: prevalence, risk factors and long-term reproductive outcome. Hum Reprod Update. 2014 Mar-Apr;20(2):262-78. doi: 10.1093/humupd/dmt045. Epub 2013 Sep 29. PMID 24082042
- [Background] Salzani A, Yela DA, Gabiatti JR, Bedone AJ, Monteiro IM. Prevalence of uterine synechia after abortion evacuation curettage. Sao Paulo Med J. 2007 Sep 6;125(5):261-4. doi: 10.1590/s1516-31802007000500002. PMID 18094891